CLINICAL TRIAL: NCT05519631
Title: Correlates Between EEG Microstates and Clinical Characteristics of People With Stroke
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Federal University of Paraíba (Other)
Responsible Party: Principal Investigator, Suellen Andrade, Principal Investigator, Federal University of Paraíba
Other Study IDs: microstates_stroke_Obs
Record Dates: First submitted 2022-08-04; First posted 2022-08-29 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Stroke; Electroencephalogram
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- subacute stroke: Participants were evaluated for clinical outcome before the electroencephalogram examination. They were evaluated with the National Institute of Health Stroke Scale (NIHSS) to quantify the severity and magnitude of neurological deficit after stroke and by the Montreal Cognitive Assessment (MoCA) to assess cognitive function.
  Interventions: Other: electroencephalogram
- chronic stroke: Participants were evaluated for clinical outcome before the electroencephalogram examination. They were evaluated with the National Institute of Health Stroke Scale (NIHSS) to quantify the severity and magnitude of neurological deficit after stroke and by the Montreal Cognitive Assessment (MoCA) to assess cognitive function.
  Interventions: Other: electroencephalogram
- healthy: Only the EEG will be collected
  Interventions: Other: electroencephalogram

INTERVENTIONS:
Other: electroencephalogram — The EEG is the recording of electrical activity in the brain in different regions of the cortex. The capture of electrical signals is performed by attaching electrodes to the surface of the scalp. As the EEG signal has an amplitude in microvolts (µVpp) it is necessary to use amplifiers, leaving the signal possible to be registered. The electrode-electrolyte interface is very important and must be able to provide a good connection between the skin and the conductive material of the electrode, otherwise the EEG signal, in addition to being contaminated by noise, may suffer distortion.

SUMMARY:
Stroke has been considered one of the main causes of long-term disability in the adult population, and is no longer considered a disease of the elderly, since 2/3 of all strokes occur among people under 70 years of age. According to the Ministry of Health, stroke is responsible for 40% of early retirements, being one of the most important causes of mortality in Brazil. The electroencephalogram (EEG) has been shown to be a very useful tool in the study of functional status and for the diagnosis of brain damage and disorders. It is considered a simple, non-invasive test with high temporal resolution, being a method widely used in laboratories to non-invasively monitor brain activity.

DETAILED DESCRIPTION:
Stroke has been considered one of the main causes of long-term disability in the adult population, and is no longer considered a disease of the elderly, since 2/3 of all strokes occur among people under 70 years of age. According to the Ministry of Health, stroke is responsible for 40% of early retirements, being one of the most important causes of mortality in Brazil. Stroke usually causes long-term deficits such as asymmetrical muscle weakness between limbs, impaired proprioceptive ability, sensory loss, vision problems, and spasticity. In addition, these sensorimotor deficits interfere with various functions of the lower limbs, including balance, postural control, and gait ability, affecting their quality of life. The electroencephalogram (EEG) has been shown to be a very useful tool in the study of functional status and for the diagnosis of brain damage and disorders. It is considered a simple, non-invasive test with high temporal resolution, being a method widely used in laboratories to non-invasively monitor brain activity. Microstates reflect short periods (~100 ms) of nearly stable brain states evolving over time, resulting from the synchronous and coordinated activity of brain networks. The aim of this study is to observe whether EEG microstates have correlations with clinical characteristics of people with stroke.

ELIGIBILITY:
Inclusion Criteria:

* people over 18 years of age, regardless of sex and with a stroke confirmed by computed tomography or magnetic resonance imaging.

Exclusion Criteria:

* have other associated neurological pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The sample consisted of 45 people, 15 individuals with subacute stroke, 15 individuals with chronic stroke and 15 healthy controls, selected for convenience. Stroke subjects were recruited through personal invitations from individuals admitted to a hospital's neurology outpatient clinic.
  Individuals matched by sex and age, with no history of neurological or psychiatric diseases, were recruited to the control group.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2023-01-30 (Actual); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-09-20 (Estimated)

PRIMARY OUTCOMES:
eeg microstates | Immediately after evaluation
  We will determine the number of topographic maps using a pre-determined criterion of the four "classical" maps (A, B, C and D) and classify the continuous EEG data according to the topographic map with which a given stretch has the highest correlation.

SECONDARY OUTCOMES:
Relationship between microstates and injury severity | Immediately after evaluation
  They were evaluated with the National Institute of Health Stroke Scale (NIHSS) to quantify the severity and magnitude of the neurological deficit after the stroke.
Relationship between microstates and cognitive function | Immediately after evaluation
  assessment of cognitive function - Montreal Cognitive Assessment (MoCA)

CONTACTS AND LOCATIONS:
Overall Officials: Suellen Andrade, Dra, Principal Investigator — Federal University of Paraiba
Locations (1):
- Aging and Neuroscience Studies Laboratory, João Pessoa, Brazil

IPD SHARING:
Plan to Share IPD: No